CLINICAL TRIAL: NCT04840836
Title: A Prospective Observational Study of the Implementation of Telehealth-Supported LARC Provision in School-Based Health Centers
Brief Title: Study of the Implementation of Telehealth-Supported LARC Provision in School-Based Health Centers
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAT6596
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Long Acting Reversible Contraception; Contraception Behavior
Keywords: LARC
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telehealth-supported LARC provision: Patients who receive care at the SBHC provide informed consent for care, as well as record review for quality assurance purposes. Analyses will include female patients who have a "reproductive health visit," which includes contraceptive counseling, contraceptive management, or contraceptive method initiation, during the study period. Patients who have a telehealth consultation with a SBHC medical provider for LARC services (conservatively estimated n=113) will be considered enrolled patients once the data are extracted from the electronic health record (EHR) system.
  Interventions: Behavioral: Telehealth-supported LARC provision

INTERVENTIONS:
Behavioral: Telehealth-supported LARC provision — Provision of LARC in routine care will include a hybrid model of telehealth-supported long-acting reversible contraception (LARC) service provision in a network of 6 school-based health centers (SBHCs) in New York City that serve adolescents and young adult high school students age 13-22 years (hereafter referred to as "adolescents").
  Other Names: LARC method

SUMMARY:
This is a prospective observational cohort study that will include SBHC patients at the 6 participating SBHCs who receive a reproductive health visit as part of their care in a setting where telehealth-supported care is available. Information will be collected during patient interviews in the follow-up observation period regarding LARC initiation, satisfaction and continuation.

Aim 1. Quantify uptake of LARC (contraceptive implant, IUD) within the SBHC network following implementation of telehealth-supported LARC provision.

Aim 2: Describe the implementation of telehealth-supported long-acting reversible contraception (LARC) service provision in school-based health centers (SBHCs) using mixed methods.

Aim 3: Quantify LARC continuation, as in absolute continuation rate 12 months post-initiation, with analyses also examining continuation at 6 months follow-up period, among LARC initiators within the SBHC network following implementation of telehealth-supported LARC provision.

Aim 4: Compare continuation rates across dimensions of telehealth experience.

DETAILED DESCRIPTION:
Long acting reversible contraceptives (LARCs) are safe and effective for adolescents, but low rates of use among this population and early discontinuation due to method dissatisfaction limits their potential to reduce unintended pregnancy. Reducing barriers for obtaining LARCs by adolescents who want to use them is key in reducing risk of unintended pregnancy. Data will be collected from patients who are receiving same-day LARC as a part of their normal care via telehealth services in school-based health centers (SBHCs). This implementation model, therefore, has the potential for replication and scale-up with wide reach. The findings from this study, given the SBHC setting, have the potential to inform and improve LARC service delivery for adolescents far beyond New York City and the SBHC setting.

ELIGIBILITY:
Inclusion Criteria:

* an enrolled patient at the participating SBHC
* age 13-22 years
* female
* had a visit at the SBHC during the study period that is coded as a "reproductive health visit" including contraceptive counseling, contraceptive management, and contraceptive method initiation

Exclusion Criteria (specifically for Aims 2 and 3):

* are younger than age 13 years
* are older than age 22
* are not an enrolled patient of the participating SBHCs
* did not initiate a LARC method
* are a person without a uterus
* are unable to read, speak, and understand either English or Spanish

Ages: 13 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Based on SBHC clinical data from the full academic year (2018-19), it is estimated that, over the 12 month cohort there will be 113 telehealth consultations, defined as a visit in which an appointment is scheduled to initiate a LARC methods (Aim 1), and 102 LARC insertions (Aim 2). The SBHC patient population, as a whole, is 69% Hispanic and 26% Black (not mutually exclusive), with an average age of 16 years.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Garbers, PhD, Principal Investigator — Associate Professor of Population & Family Health
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: device initiations
Groups:
- Telehealth-supported LARC Provision: Patients who receive care at the SBHC provide informed consent for care, as well as record review for quality assurance purposes. Analyses will include female patients who have a "reproductive health visit," which includes contraceptive counseling, contraceptive management, or contraceptive method initiation, during the study period. Patients who have a telehealth consultation with a SBHC medical provider for LARC services will be considered enrolled patients once the data are extracted from the EHR.
  Telehealth-supported LARC provision: Provision of LARC in routine care will include a hybrid model of telehealth-supported long-acting reversible contraception (LARC) service provision in a network of 6 school-based health centers (SBHCs) in New York City that serve adolescents and young adult high school students age 13-22 years (hereafter referred to as "adolescents").
Period: Overall Study
Arm/Group | Telehealth-supported LARC Provision
Started | 75; 77 device initiations
Completed | 75; 77 device initiations
Not Completed | 0; 0 device initiations

BASELINE CHARACTERISTICS:
Groups:
- Telehealth-supported LARC Provision: Patients who receive care at the SBHC provide informed consent for care, as well as record review for quality assurance purposes. Analyses will include female patients who have a "reproductive health visit," which includes contraceptive counseling, contraceptive management, or contraceptive method initiation, during the study period. Patients who have a telehealth consultation with a SBHC medical provider for LARC services (conservatively estimated n=113) will be considered enrolled patients once the data are extracted from the EHR.
  Telehealth-supported LARC provision: Provision of LARC in routine care will include a hybrid model of telehealth-supported long-acting reversible contraception (LARC) service provision in a network of 6 school-based health centers (SBHCs) in New York City that serve adolescents and young adult high school students age 13-22 years (hereafter referred to as "adolescents").
Arm/Group | Telehealth-supported LARC Provision
Number analyzed (Participants) | 75
Age, Continuous [Mean (Full Range); unit: years] | 16.65 [14 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 7
  More than one race | 26
  Unknown or Not Reported | 31
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Telehealth and Non-Telehealth LARC Device Initiations Within the SBHC Network
Description: Among all patients who had a visit for contraceptive counseling, quantify the number of telehealth LARC consultations and LARC initiations overall, and compare by LARC type (contraceptive implant vs. IUD) using data collected from patient interviews.
Time Frame: Up to 20 months
Measure: Count of Units; unit: device initiations
Units Other Than Participants: device initiations
Arm/Group | Telehealth-supported LARC Provision
Number analyzed (Participants) | 75
Number analyzed (device initiations) | 77
device initiations
  Telehealth visit | 4
  No telehealth visit | 73

2. Primary Outcome: Percentage of Patients Reported Being Satisfied With Telehealth-supported Care
Description: A qualitative interview and a quantitative survey will be used to assess LARC patients' experience and satisfaction with telehealth-supported care. Patients will be assessed by investigator as satisfied or not satisfied based on their responses.
Time Frame: Up to 20 months
Measure: Count of Units; unit: Device initiator survey respondent
Units Other Than Participants: Device initiator survey respondent
Arm/Group | Telehealth-supported LARC Provision
Number analyzed (Participants) | 43
Number analyzed (Device initiator survey respondent) | 45
Device initiator survey respondent
  Very satisfied with post-initiation visit | 33
  Somewhat satisfied with post-initiation visit | 3
  Somewhat dissatisfied with post-initiation visit | 0
  Very dissatisfied with post-initiation visit | 0
  Did not respond | 9

3. Primary Outcome: LARC Continuation Rate Over a Follow-up Period Among LARC Initiators Within the SBHC Network Following Implementation of Telehealth-supported LARC Provision
Description: Using EHR data for all patients who initiated LARC, investigator will use Kaplan-Meier survival curves to assess LARC discontinuation overall. Continuation rate will be expressed as a percentage at 6 months post-initiation, and using Kaplan-Meier curves to model discontinuation.
Time Frame: At 6 months post LARC initiation
Population: Only distinct initiators are included in this analysis. The 2 patients who initiated more than one LARC method were only counted once here; one patient had two IUD insertions, the other had IUD followed by contraceptive implant. The patient is included with their initial method in this analysis.
Measure: Median (95% Confidence Interval); unit: percent
Units Other Than Participants: device initiations
Arm/Group | Telehealth-supported LARC Provision
Number analyzed (Participants) | 75
Number analyzed (device initiations) | 75
percent
  Overall | 79.3 [69.0 to 91.1]
  Contraceptive implant: number analyzed (Participants) | 52
  Contraceptive implant: number analyzed (device initiations) | 52
  Contraceptive implant | 80.7 [68.7 to 94.8]
  IUD: number analyzed (Participants) | 23
  IUD: number analyzed (device initiations) | 23
  IUD | 76.7 [59.1 to 99.6]

4. Other Pre Specified Outcome: Continuation Rate Across Dimensions of Telehealth Experience
Description: Merging electronic health record (EHR) data on method continuation with baseline survey data on the telehealth experience, we will compare, using Cox proportional hazard models, continuation (overall and within LARC type): by telehealth experience (e.g. satisfaction with telehealth).
Time Frame: Up to 20 months
Population: Due to low number of LARC initiations, there was insufficient statistic power to detect differences in continuation. The data therefore cannot be analyzed.
Arm/Group | Telehealth-supported LARC Provision
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 20 months
Arm/Group | Telehealth-supported LARC Provision
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04840836/Prot_SAP_000.pdf